CLINICAL TRIAL: NCT03882684
Title: Role of Genomic Imprinting in Cancer Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Alliance Against Lung Cancer (Other)
Collaborators: LiSen Imprinting Diagnostic Inc. (Unknown)
Responsible Party: Principal Investigator, Bai Chunxue, Chair, Chinese Alliance Against Lung Cancer
Other Study IDs: CAALC-005-LiSen
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Early Diagnosis; Cancer; Biomarker; Genomic Imprinting
MeSH Terms: conditions — Disease; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study collects biopsies samples including but not limited to bronchoscopy biopsy, bronchial lavage fluid, fine needle aspiration, cystoscopy biopsy, urine samples, colonoscopy biopsy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients: The patients receive the surgery according to the indication of surgery. The diagnosis is confirmed by pathology of removed tissue. The result of imprinting detection are used as cancer group.
  Interventions: Diagnostic Test: In-situ imprinting detection
- Benign tumor and other disease patients: Patients ruled out the possibility of malignancy according to biopsy pathology are used as negative control.
  Interventions: Diagnostic Test: In-situ imprinting detection

INTERVENTIONS:
Diagnostic Test: In-situ imprinting detection — The loss of imprinting (LOI) and copy number variation (CNV) from biopsies will be tested by LiSen in-situ imprinting detection.

SUMMARY:
The current research focus for cancer diagonosis is classical genetics, named "driving genes". However, not all cancer patients have typical genetic alterations, especially at early stage. In the past dacades, accumulating evidences have revealed that more than 80% diseases are closely related to epigenetic changes. The normally silenced copy of imprinted genes are reactivated at early stage of cancers, and finally proceed to copy number variation. This study will screen for a panel of imprinted genes and build quantitative models to assist the diagnosis of multiple cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with suspicious cancer by ultrasound, CT or endoscope.
* Biopsy samples available.
* Male or female patients aged ≥ 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Age under 18 years.
* Severe cardiovascular diseases.
* Central nervous system diseases.
* Mental disorder.
* Pregnant.
* Individuals unwilling to sign the IRB-approved consent form and unwilling to follow the protocol to submit the serial urine for test after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with suspicious cancer in Zhongshan Hospital from July 2017 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of imprinting cancer early detection | In the middle of the study, an average of 15 months
  Number of patients "declared positive" with the imprinting early detection among the patients suffered from cancer
Specificity of imprinting cancer early detection | In the middle of the study, an average of 15 months
  Number of patients "declared negative" with the imprinting early detection among the patients who are with benign tumors or other diseases

SECONDARY OUTCOMES:
Comparison of the sensitivity of the imprinting detection versus cytopathology | In the middle of the study, an average of 15 months
  Number of patients "declared positive" with the imprinting early detection versus patients "declared positive" with the cytopathology
Comparison of the specificity of the imprinting detection versus cytopathology | In the middle of the study, an average of 15 months
  Number of patients "declared negative" with the imprinting early detection versus patients "declared negative" with the cytopathology

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feinberg AP. The Key Role of Epigenetics in Human Disease Prevention and Mitigation. N Engl J Med. 2018 Apr 5;378(14):1323-1334. doi: 10.1056/NEJMra1402513. No abstract available. PMID 29617578
- [Background] Jelinic P, Shaw P. Loss of imprinting and cancer. J Pathol. 2007 Feb;211(3):261-8. doi: 10.1002/path.2116. PMID 17177177
- [Background] Haig D. Maternal-fetal conflict, genomic imprinting and mammalian vulnerabilities to cancer. Philos Trans R Soc Lond B Biol Sci. 2015 Jul 19;370(1673):20140178. doi: 10.1098/rstb.2014.0178. PMID 26056362
- [Background] Nilendu P, Sharma NK. Epigenomic Hard Drive Imprinting: A Hidden Code Beyond the Biological Death of Cancer Patients. J Cancer Prev. 2017 Dec;22(4):211-218. doi: 10.15430/JCP.2017.22.4.211. Epub 2017 Dec 30. PMID 29302578
- [Background] Uribe-Lewis S, Woodfine K, Stojic L, Murrell A. Molecular mechanisms of genomic imprinting and clinical implications for cancer. Expert Rev Mol Med. 2011 Jan 25;13:e2. doi: 10.1017/S1462399410001717. PMID 21262060